CLINICAL TRIAL: NCT05102461
Title: Monitoring the Effects of Probiotic Supplementation in Immunocompromised Kidney Transplanted Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It wasn't approved for using Florajen as a dietary supplement and the supplier did not support the application for an IND
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1424802
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2020-08

CONDITIONS: Diarrhea Caused by Drug; Dysbiosis
Keywords: Post-Transplant Diarrhea; Gastrointestinal Symptoms; Immunosuppression Acquired Diarrhea (IAD); Probiotic Supplementation
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled study in SUNY Upstate University Hospital's Department of Surgery/Transplant Division. The total number of subjects enrolled will be 70 for both arms - placebo, 35 and treatment, 35. In order to eliminate bias, subjects will be randomized into two groups (treatment and placebo) using block randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A statistician will provide the randomization scheme to the unblinded pharmacy research staff who will carry out the process. The chance that subjects will receive Florajen Digestion or the placebo will be 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized in the Placebo Arm will take one placebo capsule daily. Each capsule will also contain 32 mg of riboflavin as a tracer substance for tracking compliance.
  Interventions: Dietary Supplement: Placebo Supplementation
- Treatment (Active Comparator): Subjects randomized in the Treatment Arm will take one placebo capsule daily. One Florajen Digestion capsule contains 15 billion live cultures of Lactobacillus acidophilus (7.5 billion), Bifodobacterium lactis (6.0 billion), and Bifidobacterium longum (1.5 billion). Each capsule will also contain 32 mg of riboflavin as a tracer substance for tracking compliance.
  Interventions: Dietary Supplement: Florajen Digestion Supplementation

INTERVENTIONS:
Dietary Supplement: Florajen Digestion Supplementation — Subjects will take the placebo starting from Week 3 post-transplant until 180 days after transplant. Compliance will be measured through the return of empty packs and urinalysis for riboflavin during follow-up visits in clinic.
  Arms: Treatment
Dietary Supplement: Placebo Supplementation — Subjects will take Florajen Digestion starting from Week 3 post-transplant until 180 days after transplant. Compliance will be measured through the return of empty packs and urinalysis for riboflavin during follow-up visits in clinic.
  Arms: Placebo

SUMMARY:
In order to protect their new renal graft, post-transplant patients follow a rigorous immunosuppressive therapy combined with prophylactic antibiotic treatment. Kidney transplant recipients are prescribed long-term immunosuppression maintenance regimens that are the prophylaxis of organ rejection. The most frequently used are calcineurin inhibitors (tacrolimus or cyclosporine) combined with glucocorticoids (methylprednisolone, prednisone) and antiproliferative agents (mycophenolate mofetil, azathioprine). However, the use of immunosuppressive medication in transplanted patients have well-documented limitations. Recent studies reported major changes in microbiota composition as a result of immunosuppression use. A large majority of transplant patients develops severe GI problems, with the most common complication being post-transplant diarrhea. Several studies have assessed and confirmed negative effects of post-transplant diarrhea. According to (3, 4), post-transplant diarrhea affects 1 in 5 patients in the first year after kidney transplantation and is associated with decreased quality of life, allograft failure, and even death.

DETAILED DESCRIPTION:
Challenges faced by patients after kidney transplantation prompted providers to look for additional strategies to improve their quality of life and decrease graft risks. In daily practice, investigators noted that a good percentage of transplant patients develops gastrointestinal (GI) symptoms, particularly diarrhea. In literature, this is known as Immunosuppression Acquired Diarrhea (IAD). These episodes are especially distressing and usually lead to immunosuppressive medication being reduced in dose or stopped. As a result of these actions, transplant patients become exposed to rejection, graft loss, and even death. Considering how the microbiota is altered during the post-transplant medication regimen, restoring the gut balance through the administration of probiotics presents a suitable solution. The proposed research would help increase knowledge on the beneficial effects and safety of probiotics in post-transplant patients.

Diarrhea is a very common and severe complication in post-transplant patients. In the majority of the cases, it is categorized as unspecified noninfectious diarrhea (1, 3). Transplant physicians associate it with immunosuppressive drugs such as mycophenolate mofetil (MMF) (7) and other agents such as tacrolimus, azathioprine, and adrenal corticosteroids that are the prophylaxis of organ rejection in patients receiving allogenic renal transplants.

The most common strategy to reduce post-transplant noninfectious diarrhea is the reduction of MMF dosing (4). Many times, the diarrhea events are so severe that the recipient's immunosuppressive medications are tapered, changed or stopped. As a result, patients become at risk of early acute rejection and graft loss.

There is a large body of literature that offers information about the etiology of diarrhea for these patients. The main cause is an alteration in microbiota composition - a condition known as dysbiosis. Offering great insight, Swarat et al., (8) wrote, "the microbiota is able to induce disease (10, 12) and also able to regulate immunity or tolerance. An imbalance between pathogenic and protective microbes characterizes dysbiosis, a perturbation in the normal composition of commensal microbiota". In the post-transplant patient population, the immunosuppressive regimen and use of prophylactic antimicrobial treatments create new post-transplant microbiota communities. In literature, dysbiosis is associated with clinical conditions and systematic inflammation.

Four main phyla found in the GI tract are known to contribute to human health and disease: Firmicutes, Bacteroidetes, Actinobacteria, and Proteobacteria, with the majority of species being non-pathogenic [13]. These commensal microbes play an important role in immune regulation, nutrition, and maintenance of host barriers against pathogens [14, 15]. It was reported that during diarrhea episodes (dysbiosis) in post-transplant patients, there is an increase in Proteobacteria and a decrease in Bacteroides, Ruminococcus, Coprococcus, and Dorea.

Although there are clinical trials offering information about microbiota composition in patients with diarrhea, there is not much information that links it to probiotic use after kidney transplantation.

The main objectives of this clinical trial are:

1. To investigate if daily use of low dose probiotics is effective in alleviating symptoms of diarrhea as well as lowering pro-inflammatory and inflammatory biomarkers and increasing anti-inflammatory biomarkers in renal transplant recipients.
2. To characterize microbiota in subjects with and without diarrhea and determine if there is any correlation between microbiota content and pro-inflammatory, inflammatory, and anti-inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a living or deceased donor kidney transplant
* Maintenance of a therapeutic dose of Mycophenolate Mofetil (MMF) and Tacrolimus after transplant
* No other gastrointestinal issues

Exclusion Criteria:

* Currently pregnant and lactating
* Has been receiving probiotics supplementation other than the study designated formula
* Participation in a different clinical trial
* Positive infection of Clostridium difficile and/or rotavirus as analyzed by stool culture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To investigate if daily use of low dose probiotics is effective in alleviating symptoms of diarrhea in post-transplant subjects | 180 days
  Does a small dose of daily probiotic supplementation improve the quality of life for kidney transplanted patients? Reduction and correction of diarrhea will be measured by <3 well-formed daily bowel movements, <200 grams of daily stool, and <75-85% fecal water content.
Correlation of probiotic use with pro-inflammatory, inflammatory, and anti-inflammatory biomarkers | 180 days
  Does probiotic supplementation lower pro-inflammatory and inflammatory biomarkers while increasing anti-inflammatory biomarkers in renal transplant recipients?
  Pro-inflammatory cytokines: Interleukin (IL)-1, IL-12, IL-13, IL-17A, tumor necrosis factor (TNF)-α and interferon (INF)-γ Inflammatory and anti-inflammatory cytokines: IL-6 and IL-4, and IL-10, respectively. Reduction and increments will be measured by the lowering or increasing of serum cytokine by 20% from baseline

SECONDARY OUTCOMES:
To characterize microbiota in subjects with and without diarrhea | 180 days
  Positive correlations will exist between "good" fecal microbiota content shifts and reductions in serum pro-inflammatory cytokine values. "Good" fecal microbiota shifts are defined as increases in Firmicutes, Bacteroides, Ruminococcus, Coprococcus, and Dorea and decreases in Protobacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Laftavi, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Lee JR, Magruder M, Zhang L, Westblade LF, Satlin MJ, Robertson A, Edusei E, Crawford C, Ling L, Taur Y, Schluter J, Lubetzky M, Dadhania D, Pamer E, Suthanthiran M. Gut microbiota dysbiosis and diarrhea in kidney transplant recipients. Am J Transplant. 2019 Feb;19(2):488-500. doi: 10.1111/ajt.14974. Epub 2018 Jul 21. PMID 29920927
- [Background] Ekberg H, Kyllonen L, Madsen S, Grave G, Solbu D, Holdaas H. Increased prevalence of gastrointestinal symptoms associated with impaired quality of life in renal transplant recipients. Transplantation. 2007 Feb 15;83(3):282-9. doi: 10.1097/01.tp.0000251923.14697.f5. PMID 17297402
- [Background] Bunnapradist S, Neri L, Wong W, Lentine KL, Burroughs TE, Pinsky BW, Takemoto SK, Schnitzler MA. Incidence and risk factors for diarrhea following kidney transplantation and association with graft loss and mortality. Am J Kidney Dis. 2008 Mar;51(3):478-86. doi: 10.1053/j.ajkd.2007.11.013. PMID 18295064